CLINICAL TRIAL: NCT06320444
Title: Developing Novel Non-invasive Electrophysiological Biomarkers of Dysfunction in Spinal and Cortical Pathways and Sensorimotor Impairments in Motor Neurone Disease
Brief Title: Non-invasive Spinal, Cortical, and Sensorimotor Biomarkers in Motor Neurone Disease
Status: Recruiting | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Motor Neurone Disease Association, UK (Unknown); Irish Research Council, IE (Unknown); Health Research Board, IE (Unknown); Research Motor Neurone, IE (Unknown); Thierry Latran Foundation, FR (Unknown); ALS Association, USA (Unknown)
Responsible Party: Principal Investigator, Orla Hardiman, Professor of Neurology, University of Dublin, Trinity College
Other Study IDs: CRFSJ0297
Record Dates: First submitted 2022-12-19; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis; Motor Neuron Disease Progressive Spinal Muscle Atrophy; Primary Lateral Sclerosis; Multiple Sclerosis; Postpoliomyelitis Syndrome
Keywords: Electroencephalography (EEG); Peripheral Nerve Stimulation; Vibration-Induced Stimulation; Neurodegeneration; Electrophysiology; Biomarkers; Neuromuscular Physiology; Spinal Connectivity
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Multiple Sclerosis; Postpoliomyelitis Syndrome; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Controls: Individuals from the Irish population with no psychiatric, psychological, neurological or muscular disease diagnosis
  Interventions: Procedure: 232 Electrode Electrophysiology (EEG-ECG-EMG-EXG)
- Amyotrophic lateral sclerosis Patients
  Interventions: Procedure: 232 Electrode Electrophysiology (EEG-ECG-EMG-EXG)
- Multiple Sclerosis patients
  Interventions: Procedure: 232 Electrode Electrophysiology (EEG-ECG-EMG-EXG)
- Postpoliomyelitis syndrome patients
  Interventions: Procedure: 232 Electrode Electrophysiology (EEG-ECG-EMG-EXG)
- Muscular Atrophy patients
  Interventions: Procedure: 232 Electrode Electrophysiology (EEG-ECG-EMG-EXG)

INTERVENTIONS:
Procedure: 232 Electrode Electrophysiology (EEG-ECG-EMG-EXG) — Noninvasive 232 Channel Electrode Electrophysiological signals (EEG-ECG-EMG-EXG) will be recorded from electrodes placed in a montage over the scalp, neck,and upper back along with muscles located on the hand. These signals will be recorded while resting or performing voluntary task.
  Other Intervention: The 232 electrode noninvasive electrophysiological data will be recorded in response to non-invasive peripheral nerve stimulation or vibration induced stimulation.
  These sessions are designed to engage specific cortical motor networks of interest for evaluating sensorimotor networks. (Cognitive, behavioural, motor, spinal, and sensory)
  Other Names: Peripheral Nerve Stimulation; Vibration Induced Stimulation

SUMMARY:
Substantial variability exists in the onset, and rate of degeneration across individuals with Motor Neurone Disease (MND) or Amyotrophic Lateral Sclerosis (ALS). This variability requires biomarkers that accurately classify and reliably track clinical subtypes as the disease progresses. Degeneration occurs in the brain and spinal cord, however, non-invasive diagnosis of spinal cord function remains highly challenging due to its unique alignment in spine. Disruption of complex spinal and cortical circuits that transmit and process neural signals for position sense and movement has not been adequately captured in the neurophysiological profiling of ALS patients. The overarching aim of this study is to reveal and quantify the extent of change in the sensorimotor integration and its potential contribution to network disruption in ALS.

DETAILED DESCRIPTION:
Background:

Substantial variability exists in the onset, and rate of degeneration across individuals with Motor Neurone Disease (MND) or Amyotrophic Lateral Sclerosis (ALS). This variability requires biomarkers that accurately classify and reliably track clinical subtypes as the disease progresses. Degeneration occurs in the brain and spinal cord, however, non-invasive diagnosis of spinal cord function remains highly challenging due its unique alignment in the spine. Disruption of complex spinal and cortical circuits that transmit and process neural signals for position sense and movement has not been adequately captured in the neurophysiological profiling of ALS patients.

Aim:

To develop, test, and employ non-invasive techniques to explore (dys)function between motor, sensory brain, and spinal networks in ALS. The project will address if the electrical activity of the cortical-spinal network by the of use peripheral stimulation (vibration, electrical nerve stimulation) to probe and reveal the normal or abnormal communication between brain and spinal networks. It is expected to reveal novel neurophysiological signatures in ALS patients compared to healthy controls.

Study Design & Data Analysis:

Surface electrodes will be mounted over the targeted regions in conjunction with High-Density EEG and High-density Electromyography (EMG). A physical and mathematical model of the underlying sources of electric activity (source localization) will be carried out at rest, during task, and with non-invasive peripheral nerve stimulation (PNS) and TMS. A separate paradigm will augment sensorimotor communication between the primary motor cortex (M1) and the somatosensory cortex (S1). Mild vibration (5N/< 500 grams) will be applied to the wrist and/or bicep tendon transcutaneously. Vibration in conjunction with non-invasive peripheral nerve stimulation will induce transient changes (30 seconds maximum) in the intrinsic excitability of motor neurons in the spinal cord. Surface EMG will capture altered MN activity at the spinal level and the anticipated augmented communication in cortical networks (S1-M1) will be captured with EEG through connectivity analysis. Non-invasive transcranial magnetic stimulation in conjunction with vibration/nerve stimulation will be recorded to explore upper motor neurone influences on the altered intrinsic excitability of spinal motor neurons.

Data collection:

EXG-EEG-EMG and TMS/Peripheral Stimulation recordings will be conducted using a BioSemi® ActiveTwo system with 128 active sintered Ag-AgCl electrodes and headcaps (BioSemi B.V., Amsterdam, The Netherlands). The TMS system is a Brainbox DuoMAG (Brainbox Ltd., Cardif, Wales, UK) which can be used with a Digitimer peripheral stimulator.

ELIGIBILITY:
Inclusion Criteria:

-

Healthy Volunteers:

* age and gender matched to patient groups
* intact physical ability to take part in the experiment.

Patients:

* Diagnosis of ALS, PLS, PMA, SMA, Polio or MS
* capable of providing informed consent.

Exclusion Criteria:

-

Healthy Controls:

* History of neuromuscular
* neurological or active psychiatric disease disease
* history of reaction or allergy to recording environments, equipment and the recording gels.

Patients:

* presence of active psychiatric disease
* any medical condition associated with severe neuropathy (e.g. poorly controlled diabetes).
* History of reaction or allergy to recording environments, equipment and the recording gels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and patients diagnosed with ALS, MS, PLS, PMA, and SMA.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Biomarker of sensorimotor integration | Baseline to 2-years after baseline
  A viable biomarker of sensorimotor integration for reliable and early distinction between healthy people and Motor Neuron Disease patient sub-phenotypes.
  This will be achieved by comparing connectivity measures between EEG, Non-cortical CNS, and EMG electrophysiological signals. The integration will also be seen in spectral analysis measures.
Determination of the feasibility of sensorimotor signatures as reliable biomarkers of ALS | Baseline
  The sensorimotor integration and signature biomarkers achieved during outcome 1 will be correlated with the clinical scores and will be statistically tested for reliability and robustness. The effect sizes of these statistical and correlation matrices will be used to evaluate the feasibility of the signatures as reliable biomarkers for motor neuron conditions like ALS.
Non-invasive recording of the SC functional neuro-electric activity | Baseline
  Understanding the role of spinal cord (SC) in neuromuscular physiology (in both impaired and healthy individuals) and will also assist in discovering biomarkers in Brain-SC Peripheral connections. This is a perspective outcome that will be future based upon the inferences gained by the first two outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Orla Hardiman, BSc MB BCh BAO MD FRCPI FAAN, Principal Investigator — Academic Unit of Neurology, Trinity College Dublin, The University of Dublin
Locations (1):
- Academic Unit of Neurology, Trinity College Dublin, The University of Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Raw data from this study may be made available in anonymized form upon request from qualified investigators subject to the approval by the Data Protection Office (DPO) and Office of Corporate Partnership and Knowledge Exchanges (OCPKE) in Trinity College Dublin, the University of Dublin.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Due to ethical constraints and the time required for data quality checks, data will only be made available in fully anonymised format following the publication of results.